CLINICAL TRIAL: NCT03203408
Title: Efficacy of OSTENIL PLUS (Hyaluronic Acid) Versus SYNVISC-ONE in Patients With Tibiofemoral Osteoarthritis. A Randomised, Controlled, Double-blind, Parallel-group Study With a 6-month Follow-up
Brief Title: Efficacy of OSTENIL PLUS (Hyaluronic Acid) Versus SYNVISC-ONE in Patients With Tibiofemoral Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TRB Chemedica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OSTP-EUR-10-01; 2011-A00258-33 (Other: ID-RCB)
Record Dates: First submitted 2017-06-22; First posted 2017-06-29 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: This study was a multicentre, prospective, double-blind, randomised, controlled non-inferiority study in two parallel groups of patients followed up for six months.
Who Masked: Participant, Outcomes Assessor
Masking Description: To prevent the patients from knowing the nature of their treatment, the investigational products OSTENIL PLUS and SYNVISC-ONE were packed in identical neutral packs. OSTENIL PLUS and SYNVISC-ONE differ in appearance (product volume and viscosity, prefilled syringe) and were therefore readily identifiable by the investigator administering the investigational product (i.e. injecting investigator). The double-blind masking could be ensured thanks to the intervention of an observer who did not know the nature of the treatment, namely the evaluating investigator. The treatment was therefore administered blind to the evaluating investigator and the patient but not to the injecting investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OSTENIL PLUS (Experimental): A single intra-articular injection of sodium hyaluronate 40 mg/2.0 ml at Day 2, i.e. 2 days post Baseline (Day 0 = Week 0)
  Interventions: Device: OSTENIL PLUS
- SYNVISC-ONE (Active Comparator): A single intra-articular injection of hylan G-F 20 48 mg/6 ml at Day 2, i.e. 2 days post Baseline (Day 0 = Week 0)
  Interventions: Device: SYNVISC-ONE

INTERVENTIONS:
Device: OSTENIL PLUS — Injection into the joint cavity of the most painful knee
  Arms: OSTENIL PLUS
Device: SYNVISC-ONE — Injection into the joint cavity of the most painful knee
  Arms: SYNVISC-ONE

SUMMARY:
The main objective of the study was to demonstrate the non-inferiority of the efficacy of a single intra-articular injection of OSTENIL PLUS compared to that of a single intra-articular injection of the reference product SYNVISC-ONE in the treatment of symptomatic tibiofemoral osteoarthritis. The primary endpoint was the change in mean score on the WOMAC pain scales from D0 to D180.

DETAILED DESCRIPTION:
After a period of washout-out for NSAIDs, the patients received a single intra-articular injection of OSTENIL PLUS or of SYNVISC-ONE in the most painful knee. The study involved a preselection visit at D-7 and five further visits: at D0 (baseline, evaluation before intra-articular injection), at D2 ± 2 days (injection), at D30 ± 15 days, at D90 ± 15 days and C5 at D180 ± 15 days.

To enrol the patients as quickly as possible, 129 sites, i.e. general medical or rheumatology practices, were open. After verifying the inclusion and exclusion criteria, the evaluating investigators assigned a randomisation number based on the chronological order of inclusion of patients at their site. The patient was then sent to the injecting investigator so that he/she could give the injection of the product corresponding to the randomisation number.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 40-85 years;
* Primary knee osteoarthritis complying with the American College or Rheumatology criteria;
* Radiographically defined osteoarthritis: joint space narrowing and osteophyte in X-ray taken less than one year previously and modified Kellgren-Lawrence grade Ib-III;
* Symptoms on one side only, with a mean WOMAC A of ≥40 mm. If knee osteoarthritis is bilateral, a difference for that score between the contralateral knee and the selected knee should be of at least 20 mm;
* Pain present on at least 15 days in the month before inclusion;
* Failure or intolerance of first line analgesics and NSAIDs;
* With health insurance;
* Understanding and following the study instructions;
* Signed the informed consent.

Exclusion Criteria:

* Knee osteoarthritis that is not symptomatic or insufficiently symptomatic;
* Bilateral symptomatic knee osteoarthritis of the same severity on both sides;
* Post-traumatic secondary knee osteoarthritis;
* Knee osteoarthritis of radiographic grade I, Ia or IV;
* Exclusively patellofemoral osteoarthritis where the symptoms are principally of patellofemoral origin (Patellar syndrome);
* Symptomatic homolateral coxarthrosis;
* Varus or valgus deformation of the selected knee (deformation axis ≥15° in X-ray);
* Inflammatory rheumatism (rheumatoid arthritis, psoriatic rheumatism, articular chondrocalcinosis, gout, Paget's disease, ankylosing spondylitis, lupus, etc.);
* History of injury to the selected knee during the 6 months before inclusion;
* Venous or lymphatic stenosis of the lower limb;
* Femoral or sciatic nerve root pain of the lower limb to be tested;
* Tendinopathy (e.g. hip periarthritis);
* Treatment with intra-articular hyaluronic acid in the selected knee during the 6 months before inclusion;
* Intra-articular injection of corticosteroids in the selected knee during the 2 months before inclusion;
* Treatment with symptomatic slow-acting drugs for osteoarthritis and/or dietary supplements for osteoarthritis (chondroitin sulphate, diacerein, avocado and soybean unsaponifiables, oxaceprol, copper granions, glucosamine) which had been started less than 3 months previously or whose dose had been changed during the last 3 months before inclusion;
* Total knee replacement of the selected knee;
* Surgery of the other knee or of the hip or any other surgery scheduled during the period of the study;
* History of any surgical intervention, arthroscopy, osteotomy, etc. in the year before inclusion;
* Obesity: body mass index ≥30 kg/m2;
* History of autoimmune disease;
* Severe condition likely to interfere with the evaluation, such as neoplasia, malignant blood disease, kidney disease, liver disease or severe infection;
* Very marked hydrarthrosis (requiring puncture) at the time of inclusion;
* Wound or skin condition of the selected knee;
* Anticoagulant treatment with heparin or warfarin (platelet antiaggregants such as ASPIRIN ≤325 mg/d, ticlopidine or clopidogrel were allowed);
* Known hypersensitivity to hyaluronic acid and/or to avian proteins and/or paracetamol;
* Known hypersensitivity to mannitol;
* Participation in a clinical research study within the previous 3 months;
* Pregnancy, breast-feeding.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2011-06-21 (Actual); Primary Completion 2012-11-22 (Actual); Study Completion 2012-11-22 (Actual)

PRIMARY OUTCOMES:
Change in WOMAC A | Day 0 to Day 180
  Change from baseline in the pain subscore (section A) of the WOMAC score

SECONDARY OUTCOMES:
Lequesne algofunctional index | Day 0 to Day 180
  Index assessing the severity of osteoarthritis
WOMAC B | Day 0 to Day 180
  Stiffness subscore (section B) of the WOMAC score
WOMAC C | Day 0 to Day 180
  Function subscore (section C) of the WOMAC score
Patient's overall status score in relation to his/her knee osteoarthritis | Day 0 to Day 180
  Visual analogue scale assessed by the patient
Assessment of overall treatment efficacy by the patient | Day 30 to Day 180
  5-point scale (1 = very good; 2 = good; 3 = moderate; 4 = poor; 5 = very poor)
Assessment of overall treatment efficacy by the investigator | Day 30 to Day 180
  5-point scale (1 = very good; 2 = good; 3 = moderate; 4 = poor; 5 = very poor)

OTHER OUTCOMES:
Incidence of all adverse events | Day 0 to Day 180
  Recording of all adverse events and changes in concomitant treatments
Incidence of local adverse reactions | Day 30
  Recording of adverse manifestations such as post-injection pain, inflammatory reaction, presence of hydrarthrosis, presence of acute pseudoseptic or septic arthritis
Assessment of local treatment tolerability by the patient | Day 30
  5-point scale scale (1 = very good, 2 = good, 3= moderate, 4 = poor, 5 = very poor)
Assessment of local treatment tolerability by the investigator | Day 30
  5-point scale scale (1 = very good, 2 = good, 3= moderate, 4 = poor, 5 = very poor)
Assessment of overall treatment tolerability by the investigator | Day 30 to Day 180
  5-point scale (1 = very good; 2 = good; 3 = moderate; 4 = poor; 5 = very poor)
Assessment of overall treatment tolerability by the patient | Day 30 to Day 180
  5-point scale (1 = very good; 2 = good; 3 = moderate; 4 = poor; 5 = very poor)

CONTACTS AND LOCATIONS:
Overall Officials: Renée Liliane Dreiser, Dr, Study Chair — APHP Bichat-Claude Bernard, Paris, France; Bernard Avouac, Dr, Study Chair — APHP Henri Mondor, Creteil, France; Thomas Bardin, Prof., Principal Investigator — APHP Lariboisière, Paris, France

IPD SHARING:
Plan to Share IPD: No